CLINICAL TRIAL: NCT03726190
Title: Clinical and Radiological Outcomes of Oblique Lateral Lumbar Interbody Fusion
Status: Suspended | Type: Observational
Sponsor: Tristate Brain and Spine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 201801
Record Dates: First submitted 2018-10-27; First posted 2018-10-31 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis; Lumbar Disc Herniation
Keywords: Degenerative Disk Disease; Lumbar Fusion; Minimally Invasive Surgery; Lumbar Disk Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OLLIF: Patients who underwent Oblique Lateral Lumbar Interbody Fusion
  Interventions: Procedure: Oblique Lateral Lumbar Fusion

INTERVENTIONS:
Procedure: Oblique Lateral Lumbar Fusion — Oblique lateral lumbar interbody fusion (OLLIF) is a lumbar spinal fusion. OLLIF is performed with the patient in the prone position and employs an oblique lateral approach that enables the instrumentation to pass through Kambin's triangle which is defined as the space between the exiting nerve, the superior border of the caudal vertebra, and the superior articulating process of the inferior facet. This approach may be performed without direct visualization, guided by electrophysiological monitoring and biplanar fluoroscopy. During the approach, a blunt probe is used to make contact with the disc, followed by a series of gentle dilations. Discectomy is performed through a 10-mm access portal. The cage is inserted under continued electrophysiological monitoring and fluoroscopy.

SUMMARY:
This study is undertaken to evaluate the outcomes of Oblique Lateral Lumbar Interbody Fusion (OLLIF). Specifically, the study seeks to measure outcomes on radiological imaging, outcomes reported by the patients on standardized questionnaires, and complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis, confirmed by imaging, of one of the following conditions: severe degenerative disc disease, spondylolisthesis, spinal stenosis, disc herniation
* Completion of a full course of conservative therapy. Conservative therapy may include physical therapy, therapeutic injections, bracing and behavioral modification.

Exclusion Criteria:

* bony obstruction of the approach
* significant spinal canal stenosis
* large facet hypertrophy
* grade II listhesis
* scoliosis with Cobb angle > 10º
* Patients who underwent procedures that were converted to open fusions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who presented to the study center and required lumbar fusion were eligible to participate in this study. The study center draws patients from Minnesota, South Dakota and North Dakota. No demographic restrictions were placed on participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient reported disability on the Oswestry Disability Index | One year after surgery
  The Oswestry Disability Index is a commonly used tool to assess disability due to low back pain. The Oswestry is assessed on a standardized questionnaire and the scale ranges from 0% to 100% disability. A lower score is considered less disability.
Fusion rate | One year after surgery
  The rate of bony fusion as determined by independent radiologists on post-operative CT scans. Radiologists will determine whether each level that was operated on was fused, or not fused.
Rate of Neuropraxia | One year after surgery
  Neuropraxia is defined as lower extremity weakness of 3/5 or below on a standard 5 point strength scale as assessed by the surgeon at one year follow-up. The scale ranges from 5 (full strength) to 0 (no muscle tone). The deficit must have newly appeared just after surgery to be considered a result of the surgery.
Rate of Nerve Root Irritation | One year after surgery
  Nerve Root Irritation is defined as lower extremity paresthesias or dysesthesias corresponding to dermatome of the level of surgery or weakness of 4/5 or above on a standard 5 point strength scale as assessed by the surgeon at one year follow-up. The scale ranges from 5 (full strength) to 0 (no muscle tone). The deficit must have newly appeared just after surgery to be considered a result of the surgery.

SECONDARY OUTCOMES:
Surgery Time | During surgery
  Skin to skin surgery time measured in minutes
Hospital stay | Immediately after surgery
  The number of nights spent in the hospital following the surgery measured in days
Blood Loss | During surgery
  The amount of blood lost during the surgery measured in milliliters.
Fluoroscopy Time | During surgery.
  The time fluoroscopy was used during surgery measured in seconds.
Rate of screw fracture | One year after surgery
  The percentage of all screws placed in the study group that is determined to have fractured on postoperative imaging. Imaging is read by independent radiologists.
Infection Rate | Immediately after surgery
  The percentage of patients that experienced a postoperative surgical site infection.
Bleeding Rate | During surgery and immediately after surgery
  The percentage of patients that experienced bleeding during surgery or immediately after surgery that required transfusion.
Patient reported pain on a 10-point pain scale | One year after surgery
  The level of pain reported by the patient on a standard 10-point pain scale. The scale goes from 0 (no pain) to 10 (worst pain imaginable)

CONTACTS AND LOCATIONS:
Locations (1):
- Tristate Brain and Spine Institute, Alexandria, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
IDP data will not be made publicly available to preserve the privacy of study participants. Requests to access our data will be considered on a case by case basis to ensure that data cannot be re-identified.